CLINICAL TRIAL: NCT05056285
Title: Pattern of Growth and Characteristics of Down Syndrome Pediatrics Patients Attending Assuit University Children Hospital
Brief Title: Pattern of Growth and Characteristics of Down Syndrome Pediatrics Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Gaber Osman, Amira Gaber Osman, Assiut University
Other Study IDs: PogacoDsppaAuch
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Down syndrome less than four years Group

SUMMARY:
Down syndrome or Down's syndrome (DS), also known as trisomy 21, is a genetic disorder caused by the presence of all or part of a third copy of chromosome 21. It is usually associated with physical growth delays, mild to moderate intellectual disability, and characteristic facial features. The parents of the affected individual are usually genetically normal. The probability increases from less than 0.1% in 20-year-old mothers to 3% in those of age 45 .

DETAILED DESCRIPTION:
People with DS may have some or all of these physical characteristics: a small chin, slanted eyes, poor muscle tone, a flat nasal bridge, a single crease of the palm, and a protruding tongue due to a small mouth and relatively large tongue. Other features include: a flat and wide face, a short neck, excessive joint flexibility, extra space between big toe and second toe, abnormal patterns on the fingertips and short fingers. Short stature is a characteristic feature of DS. Growth retardation of DS individuals starts prenatally. After birth, the growth velocity is most reduced between 6 months to 3 years . Growth charts specific for children with DS are important tools for routine medical follow-up, as well as early identification of pathological causes of growth retardation, and monitoring of growth promoting treatments. Growth charts for DS are available from different countries, for example, Italy, USA, Denmark, Sweden, Portugal, France, UK and Ireland and Saudi Arabia .

ELIGIBILITY:
Inclusion Criteria:

* All Down syndrome children attending Assuit university less than four years with or without cardiovascular.

Exclusion Criteria:

* Any Down syndrome child more than four years.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 1. Inclusion criteria:
     All Down syndrome children attending Assuit university less than four years with or without cardiovascular .
  2. Exclusion criteria:
  Any Down syndrome child more than four years. This is a descriptive case series study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The pattern of growth in Down syndrome patients | 6 months
  Descriptive case series study

REFERENCES:
- [Background] Morris JK, Mutton DE, Alberman E. Revised estimates of the maternal age specific live birth prevalence of Down's syndrome. J Med Screen. 2002;9(1):2-6. doi: 10.1136/jms.9.1.2. PMID 11943789
- [Background] Perkins JA. Overview of macroglossia and its treatment. Curr Opin Otolaryngol Head Neck Surg. 2009 Dec;17(6):460-5. doi: 10.1097/MOO.0b013e3283317f89. PMID 19713845
- [Background] Malt EA, Dahl RC, Haugsand TM, Ulvestad IH, Emilsen NM, Hansen B, Cardenas YE, Skold RO, Thorsen AT, Davidsen EM. Health and disease in adults with Down syndrome. Tidsskr Nor Laegeforen. 2013 Feb 5;133(3):290-4. doi: 10.4045/tidsskr.12.0390. English, Norwegian. PMID 23381164
- [Background] Sara VR, Gustavson KH, Anneren G, Hall K, Wetterberg L. Somatomedins in Down's syndrome. Biol Psychiatry. 1983 Jul;18(7):803-11. No abstract available. PMID 6225471
- [Background] Piro E, Pennino C, Cammarata M, Corsello G, Grenci A, Lo Giudice C, Morabito M, Piccione M, Giuffre L. Growth charts of Down syndrome in Sicily: evaluation of 382 children 0-14 years of age. Am J Med Genet Suppl. 1990;7:66-70. doi: 10.1002/ajmg.1320370712. PMID 2149977
- [Result] Patterson D. Molecular genetic analysis of Down syndrome. Hum Genet. 2009 Jul;126(1):195-214. doi: 10.1007/s00439-009-0696-8. Epub 2009 Jun 13. PMID 19526251
- [Result] Weijerman ME, de Winter JP. Clinical practice. The care of children with Down syndrome. Eur J Pediatr. 2010 Dec;169(12):1445-52. doi: 10.1007/s00431-010-1253-0. Epub 2010 Jul 15. PMID 20632187